CLINICAL TRIAL: NCT03905967
Title: Transarterial Chemoembolization With Lenvatinib Versus Lenvatinib Alone in First-line Treatment of Advanced Hepatocellular Carcinoma: a Phase III, Multicenter, Randomized Controlled Trial
Brief Title: TACE With Lenvatinib Versus Lenvatinib Alone in in First-line Treatment of Advanced HCC
Acronym: TACE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Clinical Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20190031
Record Dates: First submitted 2019-03-28; First posted 2019-04-08 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Advanced Hepatocellular Carcinoma
Keywords: Lenvatinib; Transarterial chemoembolisation
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lenvatinib + TACE (Experimental): Patients in Lenvatinib + TACE group will take oral lenvatinib within 3 days of randomization and receive TACE 1 day after oral administration of lenvatinib.
  Interventions: Procedure: TACE; Drug: Lenvatinib
- Lenvatinib (Active Comparator): Lenvatinib alone
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Procedure: TACE — TACE will be performed one day after oral administration of lenvatinib. TACE with either cTACE or DEB-TACE can be used, depending on the condition of each center.
  Arms: Lenvatinib + TACE
Drug: Lenvatinib — Lenvatinib will be taken within 3 days of randomization (dose: 8 mg qd for patients <60kg, and 12 mg qd for patients >60kg)

SUMMARY:
This trial is is an open label, multicenter, randomized controlled phase 3 clinical trial. The purpose is to compare the efficacy and safety of lenvatinib plus TACE with lenvatinib alone for advanced HCC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old;
2. Patients with primary advanced HCC (in accordance with AASLD2018 guidelines for the diagnosis of HCC), without any previous treatment;
3. There is at least one measurable lesion in the liver according to mRECIST criteria, single tumor ≤ 10.0 cm or multiple tumors and tumor burden ≤50% , with portal vein tumor embolus or with extrahepatic metastasis;
4. ECOG score 0-1;
5. Child-Pugh class A;
6. Expected survival time ≥ 3 months;
7. Blood, liver and kidney function meet the following conditions: Neutrophil count ≥ 1.5 × 10 9 /L; Platelet count ≥ 60 × 10 9 /L; Hemoglobin ≥ 90 g/L; Serum albumin ≥ 30 g/L; Bilirubin ≤ 50 umol/L; AST, ALT ≤ 5 times the upper limit of normal, ALP ≤ 4 times the upper limit of normal; Prolongation of prothrombin time not to exceed the upper limit of normal by 6 seconds; Creatinine ≤ 1.5 times the upper limit of normal

Exclusion Criteria:

1. Preoperative imaging examination revealed diffuse intrahepatic lesions or invasion, inferior vena cava or primary branch bile duct;
2. Previous history of hepatic encephalopathy, refractory ascites or gastric esophageal varices;
3. There are contraindications to TACE treatment, such as portosystemic shunt, liver flow ablation, significant atherosclerosis;
4. Brain metastases;
5. Hypersensitivity to intravenous contrast agents;
6. Pregnant or lactating women or subjects with family planning within two years;
7. With HIV, syphilis infection;
8. Accompanied by other malignant tumors or suffering from other malignancies within 5 years before enrollment;
9. Allogeneic organ transplant recipients;
10. Severe dysfunction of heart and kidney or other organs;
11. Active severe infection > grade 2 (NCI-CTC version 4);
12. Suffering from mental and psychological diseases may affect informed consent;
13. Unable to take oral medication;
14. Participated in other drug clinical trials within 12 months before enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
Overall survival | two years
  Defined as the time from randomization to death for any cause.

SECONDARY OUTCOMES:
Time to progression | two years
  Defined as the time from randomization to disease progression.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Kudo M, Finn RS, Qin S, Han KH, Ikeda K, Piscaglia F, Baron A, Park JW, Han G, Jassem J, Blanc JF, Vogel A, Komov D, Evans TRJ, Lopez C, Dutcus C, Guo M, Saito K, Kraljevic S, Tamai T, Ren M, Cheng AL. Lenvatinib versus sorafenib in first-line treatment of patients with unresectable hepatocellular carcinoma: a randomised phase 3 non-inferiority trial. Lancet. 2018 Mar 24;391(10126):1163-1173. doi: 10.1016/S0140-6736(18)30207-1. PMID 29433850
- [Background] Forner A, Reig M, Bruix J. Hepatocellular carcinoma. Lancet. 2018 Mar 31;391(10127):1301-1314. doi: 10.1016/S0140-6736(18)30010-2. Epub 2018 Jan 5. PMID 29307467
- [Background] Meyer T, Fox R, Ma YT, Ross PJ, James MW, Sturgess R, Stubbs C, Stocken DD, Wall L, Watkinson A, Hacking N, Evans TRJ, Collins P, Hubner RA, Cunningham D, Primrose JN, Johnson PJ, Palmer DH. Sorafenib in combination with transarterial chemoembolisation in patients with unresectable hepatocellular carcinoma (TACE 2): a randomised placebo-controlled, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2017 Aug;2(8):565-575. doi: 10.1016/S2468-1253(17)30156-5. Epub 2017 Jun 23. PMID 28648803
- [Background] Park JW, Kim YJ, Kim DY, Bae SH, Paik SW, Lee YJ, Kim HY, Lee HC, Han SY, Cheong JY, Kwon OS, Yeon JE, Kim BH, Hwang J. Sorafenib with or without concurrent transarterial chemoembolization in patients with advanced hepatocellular carcinoma: The phase III STAH trial. J Hepatol. 2019 Apr;70(4):684-691. doi: 10.1016/j.jhep.2018.11.029. Epub 2018 Dec 6. PMID 30529387
- [Derived] Peng Z, Fan W, Zhu B, Wang G, Sun J, Xiao C, Huang F, Tang R, Cheng Y, Huang Z, Liang Y, Fan H, Qiao L, Li F, Zhuang W, Peng B, Wang J, Li J, Kuang M. Lenvatinib Combined With Transarterial Chemoembolization as First-Line Treatment for Advanced Hepatocellular Carcinoma: A Phase III, Randomized Clinical Trial (LAUNCH). J Clin Oncol. 2023 Jan 1;41(1):117-127. doi: 10.1200/JCO.22.00392. Epub 2022 Aug 3. PMID 35921605